CLINICAL TRIAL: NCT06076252
Title: Modified Blumgart vs Conventional Blumgart Anastomosis Technique in the Treatment of Periampulltrary Carcinoma on Postoperative Pancreatic Fistula: an Open, Randomized, Parallel Controlled Clinical Study
Brief Title: Modified vs Conventional Blumgart Anastomosis of LPD for the Effects of Pancreatic Fistula of Periampullary Carcinoma
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Guangdong Medical University (Other)
Responsible Party: Principal Investigator, Guohua Liu, Principal Investigator, Affiliated Hospital of Guangdong Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PJKT2023-061
Record Dates: First submitted 2023-08-30; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-04

CONDITIONS: Ampullary Cancer; Bile Duct Cancer; Pancreas Cancer; Duodenum Cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Pancreatic Neoplasms; Duodenal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Blumgart Anastomosis of LPD (Experimental): The effect of modified Blumgart technique in the treatment of periampulltrary carcinoma on postoperative pancreatic fistula
  Interventions: Procedure: Modified Blumgart Anastomosis in LPD
- Conventional Blumgart Anastomosis of LPD (Other): The effect of Conventional Blumgart Anastomosis in the treatment of periampulltrary carcinoma on postoperative pancreatic fistula
  Interventions: Procedure: conventional Blumgart anastomosis in LPD

INTERVENTIONS:
Procedure: Modified Blumgart Anastomosis in LPD — This study is a clinical study designed by parallel control, the test group is LPD patients with modified Blumgart anastomosis and the control group is LPD patients with conventional Blumgart anastomosis
  Arms: Modified Blumgart Anastomosis of LPD
Procedure: conventional Blumgart anastomosis in LPD — This study is a clinical study designed by parallel control, the test group is LPD patients with modified Blumgart anastomosis and the control group is LPD patients with conventional Blumgart anastomosis
  Arms: Conventional Blumgart Anastomosis of LPD

SUMMARY:
The incidence rate and mortality rate of periampullary cancer at home and abroad both show an increasing trend, seriously affecting the health level of the people. Pancrecoduodenectomy (PD) is the only effective treatment for periampullary cancer. However, due to the complex technology and difficulty of PD surgery, laparoscopic pancreaticoduodenectomy (LPD) is more difficult, and the postoperative mortality can reach 5%. The important reason is the most serious complication- -pancreatic fistula. The occurrence of pancreatic fistula is related to many factors, and the most critical factor is the method and technology of pancreatico-intestinal anastomosis, so the improvement and innovation of pancreaticoco-intestinal anastomosis technology has always been a hot topic in surgical clinical research. Blumgart Pancreatic anastomosis was originally created by Professor L.H.Blumgart in the United States, and was widely used in OPD due to its low incidence of pancreatic fistula. However, the traditional Blumgart anastomosis is complicated and is not suitable for application in LPD. According to our own experience, our team simplified and improved the traditional Blumgart anastomosis to OPD, and through retrospective study, it has the advantages of reducing the incidence of pancreatic fistula. However, the application value in LPD still needs to be further discussed. Therefore, this study intends to use a prospective randomized controlled trial, using the LPD patients with traditional Blumgart pancreatecointestinal anastomosis as the control group, and the LPD patients with modified Blumgart pancreatecointestinal anastomosis as the test group, compare the clinical relevant indicators and the incidence of postoperative complications, and explore whether the application value in LPD can truly simplify the surgical procedure and ensure the lower incidence of pancreatic leakage.

DETAILED DESCRIPTION:
This study intends to use a prospective randomized controlled trial, the LPD patients with traditional Blumgart anastomosis as the control group, design the LPD patients with modified Blumgart anastomosis as the test group, by comparing the clinical correlation index and the rate of postoperative complications in LPD can truly simplify the surgical procedure and ensure the lower rate of pancreatic leakage.

The following steps will be followed:

1. Patients who met the inclusion criteria and did not meet the exclusion criteria underwent modified Blumgart anastomosis according to the randomization LPD surgery group (test group) or LPD surgery group with conventional Blumgart pancreatecreenterostomy (control group).
2. The following common LPD procedure was used in the test and control groups: ① Preoperative preparation and anesthesia mode Preoperative gastric tube, urinary tube and central venous channel; general anesthesia ② Same surgical procedure: Establishment of artificial pneumoperitoneum and operating hole anatomical exploratory specimen resection and reconstruction of digestive tract (biliary intestine kiss Combination, gastrointestinal anastomosis) drain placement.
3. In the test group, the pancreatic intestine anastomosis in the LPD Combined, the control group used conventional Blumgart pancreatestatic anastomosis.
4. Both postoperative groups were routinely given anti-infection, gastric mucosa protection, somatostatin, and nutritional supportive therapy. After the first Remove gastric tube and urinary catheter on 3 days, instructed patients to eat cold liquid food and ambulation; somatostatin was stopped on postoperative day 5, The upper abdominal CTA was reviewed, and the remaining treatment plans were formulated according to the actual situation of the patient. Postoperative numbers 1,3,5, and For 7 days, the relevant drainage indexes, daily drainage rate, drainage properties and amylase content were reviewed.
5. If the patient can be discharged with the following conditions: the general condition is good, and the normal diet and intestinal function are basically restored; Body temperature was normal and the abdominal examination showed no positive signs; relevant laboratory results were almost normal; CTA Significant abdominal effusion and other abnormalities; postoperative abdominal incision healed well.
6. After discharge, pay attention to their appetite, spirit, urine and feces, and drainage tube (discharged with drainage tube). Patients without special discomfort were returned to the hospital for review once at 1and 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

Radically resectable stage I - III low periampullary carcinoma in patients, And all met the following criteria:

1. age 18-75 years;
2. imaging (upper abdominal MRI, MRCP / CT / CTA) diagnosis of periampullary (duodenal papilla, ampulla, inferior common bile duct, pancreatic head);
3. MDT discussion of tumor invasion of large vessels (SMA, CA, CHA/SMV, PV) resectable;
4. endoscopic duodenal ultrasound diagnosis of periampullary carcinoma;
5. endoscopic biopsy pathology confirmation of carcinoma (not essential);
6. preoperative stage within T3N1;
7. no evidence of distant metastasis;
8. cardiopulmonary and liver and kidney function can tolerate surgery;
9. patients and family members can understand and willing to participate in this study, Provided the written informed consent.

Exclusion Criteria:

1. Diagnosis of malignant tumors in other sites;
2. ASA grade IV and / or ECOG physical strength status score> 2 points;
3. Patients with severe liver and kidney function, cardiopulmonary function, coagulation dysfunction or severe basic diseases who cannot tolerate surgery;
4. Have an uncontrolled preoperative infection;
5. Pregnant or lactating women;
6. A history of serious mental illness;
7. Patients with other clinical and laboratory conditions considered by the investigator are not suitable to participate in this trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
The rate of POPF | 90 Days after surgery
  The rate of Postoperative pancreatic fistula

CONTACTS AND LOCATIONS:
Overall Officials: Liu Guohua, Study Director — Affiliated Hospital of Guangdong Medical University
Locations (1):
- The Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT06076252/Prot_000.pdf